CLINICAL TRIAL: NCT03817762
Title: Respiratory Polygraphy in Children : Feasibility in Every Day Pratice in an ENT Department and Value of the Automatic Detection of Respiratory Events
Brief Title: Feasibility in Every Day Pratice in an ENT Department and Value of the Automatic Detection of Respiratory Events
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0450
Record Dates: First submitted 2018-10-04; First posted 2019-01-25 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-10

CONDITIONS: Obstructive Sleep Apnea Hypopnea Syndrome
Keywords: pediatric obstructive sleep apnea hypopnea syndrome; pediatric respiratory polygraphy; device acceptance; signal quality; automatic detection of respiratory events

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of respiratory polygraphy (RP) in children for the diagnosis of obstructive sleep apnea hypopnea syndrome (OSAHS) can be challenging: device acceptance, sensors displacement. The automatic analysis of respiratory events has never been evaluated in a pediatric population. The primary objective of this study was to determine the feasibility of pediatric RP in an ENT department routine practice. The second objective was to evaluate the reliability of the automatic signal analysis in children.

DETAILED DESCRIPTION:
Retrospective single center study of 50 children (32 boys and 18 girls, mean age 5.5 ± 2.3 years) who benefited from an overnight RP in an ENT hospitalization department between January and August 2016 for OSAS suspicion. Manual detection of respiratory events was performed by the same ENT specialist, and compared to the automatic analysis.

ELIGIBILITY:
Inclusion criteria:

* Age between 2 and 12 years
* child having performed a ventilatory polygraph for suspicion of obstructive hypopnoea apnea syndrome

Exclusion criteria:

- over 12 years old

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with clinical obstructive sleep apnea hypopnea syndrome in University Health Center
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Overall signal quality of the respiratory polygraph | 1 day
  retrospective data collection : Overall signal quality of RP (Respiratory polygraphy)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AKKARI, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France